CLINICAL TRIAL: NCT01149200
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Proof-of-Principle Study to Evaluate the Safety, Tolerability, and Efficacy of TC-6499-12 in the Treatment of Constipation Predominant IBS
Brief Title: Proof-of-Principle Study of TC-6499 in the Treatment of Constipation Predominant Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Targacept Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TC-6499-12-CLP-004
Record Dates: First submitted 2010-06-14; First posted 2010-06-23 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; IBS-C
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TC-6499 (Experimental)
  Interventions: Drug: TC-6499
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TC-6499 — 5mg enteric-coated oral hard gelatin capsule, administered twice daily
  Arms: TC-6499
Drug: Placebo — placebo as enteric-coated oral hard gelatin capsule, administered twice daily
  Arms: Placebo

SUMMARY:
Study is to assess the effectiveness of TC-6499 in the treatment of constipation predominant IBS patients over a 28-day period.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo controlled study of a maximum of 24 subjects with constipation predominant irritable bowel syndrome (IBS-C). Sixteen subjects will receive active treatment and 8 subjects will receive matching placebo. There will be a 21-day screening phase before 1st study drug administration on Day 1.

ELIGIBILITY:
Inclusion Criteria:

* Men with IBS-C (ROME III) between 18 and 65 years of age, inclusive.
* Women with IBS-C (ROME III) between 55 and 65 years of age, or 18 to 55 years of age with documentation of non-childbearing potential status (surgical sterilization or one year post last menses with elevated FSH/LV).
* All subjects should have a body mass index (BMI) between 18 and 34 kg/m2, inclusive and a body weight of not less than 45 kg.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in global IBS symptom relief score | 28 days
  Primary efficacy endpoint assessed weekly using patient's response to a global symptom relief question rating their relief of IBS symptoms over the past week compared to before study entry.

SECONDARY OUTCOMES:
Weekly number of spontaneous bowel movements (SBM) | 28 days
  The number of spontaneous bowel movements not associated with rescue medication will be assessed through patient self-reports
Severity of pain, bloating, degree of straining, and stool consistency | 28 days
  Severity of pain, bloating, degree of straining, and stool consistency will be assessed through daily patient self-reports

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, MB, ChB, Principal Investigator — Quotient Bioresearch
Locations (2):
- United Kingdom (2):
  - Quotient Clinical Ltd, Edinburgh
  - Quotient Clinical Ltd, Ruddington